CLINICAL TRIAL: NCT00787267
Title: Phase II Study of Dasatinib in Previously Treated Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Phase II Study of Dasatinib in Previously Treated Patients With Advanced NSCLC
Acronym: TOP0801
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Duke University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008303
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Results first posted 2015-01-01 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; Lung Cancer; Dasatinib; Genomics; Genomics analysis; Genomic signature
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dasatinib (Experimental): After a biopsy is done to obtain fresh frozen tumor tissue (Stage I), dasatinib is to be administered as an oral dose of 70 mg twice daily on a continuous basis for 6 weeks. Every 6 weeks radiologic exam will be done to assess response. Treatment will continue until progression of disease, intolerable toxicity or patient withdrawal.
  For Stage II, a biopsy to obtain fresh frozen tumor tissue will also be done. Depending on results from Stage I and results of biopsy, treatment with dasatinib will be determined.
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — 70 mg PO twice daily until progression. Re-assess radiographically every 6 weeks.
  Other Names: Sprycel

SUMMARY:
On this study patients will receive dasatinib, a targeted therapy, for advanced NSCLC that has progressed after previous therapy. Safety and response to dasatinib will be assessed.

Fresh frozen tumor tissue must be available for genomics analysis prior to initiating dasatinib therapy. A biopsy must be obtained after any prior chemotherapy. If fresh frozen tumor tissue is not available, a biopsy will be required to participate in this trial.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death in the United States. Twenty to seventy-five percent of patients initially treated with surgery or radiotherapy recur and become candidates for systemic therapy. Src expression has been identified in a majority of NSCLC cell lines and may be important in hypoxic growth and angiogenesis of NSCLC.

This phase II trial will investigate the activity of the oral Src inhibitor dasatinib in advanced stage NSCLC. We hypothesize that the inhibition of Src pathway with dasatinib will show anti-tumor activity in advanced NSCLC, with a tolerable safety profile.

Fresh frozen tissue is needed for the genomics analysis, thus a biopsy will be required to participate in this trial. The genomic analysis will determine if the tumor is Src-active or Src-inactive and responses to dasatinib compared. In stage I, 40 patients will be treated without prior knowledge of their tumoral Src-activity. If all stage I responses are observed in the Src-active patients, the second stage will only accrue that cohort. If all responses are observed in the Src-inactive cohort, the activity of dasatinib and genomic determination of dasatinib response will be re-evaluated. Otherwise, if during Stage I, responses are observed in both cohorts, they will be accrued separately and evaluated in a two-stage manner.

Dasatinib will be give orally twice daily and continue until progression of disease, intolerable toxicity or patient withdrawal. Imaging studies will be done pre-treatment then every 6 weeks to assess radiologic response to therapy.

Patients will be followed for 30 days after the last dose of dasatinib to assess toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Histological/cytological documented non-small cell lung cancer (NSCLC). Documentation of recurrence required if treated with surgical resection and/or external beam radiation therapy (XRT) with curative intent and now have recurrent disease.
2. Fresh tissue biopsy material for genomics analysis prior to initiating dasatinib. If prior XRT, tissue biopsy must be outside XRT field. Biopsy must be after any prior chemotherapy.
3. Prior treatment (tx) to include one of the following:

   * At least 1 prior systemic regimen (IV or oral agent) for Stage IV NSCLC or for recurrent disease.
   * Recurrence within 12 months after completion of systemic neoadjuvant/adjuvant chemotherapy for early stage NSCLC.
   * Combined modality platinum-based tx for Stage III NSCLC.
4. Prior XRT permitted if ≥1 week since completion, XRT must be <25% of bone marrow reserve.
5. At least one, non-radiated, measurable lesion (per RECIST).
6. Age ≥18 years.
7. Eastern Cooperative Oncology Group (ECOG) 0-2.
8. Adequate Organ Function:

   1. Total bilirubin < Upper limit normal (ULN)
   2. Hepatic enzymes (AST, ALT) ≤2.5x ULN
   3. Serum creatinine <1.5x ULN
   4. Hemoglobin ≥9 gm/dL
   5. Neutrophil count (ANC/AGC) ≥1500 per μL
   6. Platelets ≥100,000 per μL
   7. Prothrombin time (PT)/a Partial thromboplastin time (PTT) ≤1.5x control
9. No other serious medical or psychiatric illness.
10. Ability to take oral medication (dasatinib must be swallowed whole).
11. Women of childbearing potential must have negative serum pregnancy test ≤72 hours and not >7 days prior to starting study drug.
12. Sexually active males and females of reproductive potential must agree to use adequate method of contraception during tx and for at least 4 weeks after study drug stopped.
13. Signed, written informed consent including Health Insurance Portability and Accountability Act (HIPAA) according to institutional guidelines.

Exclusion Criteria:

1. Previous or concomitant malignancy in past 2 years other than curatively treated carcinoma in situ of cervix, or basal cell/squamous cell carcinoma of the skin.
2. Prior tx with dasatinib or other agents that inhibit Src.
3. Evidence of symptomatic pleural effusions (grade 2) unless undergo therapeutic thoracentesis as part of non-study care. Successful pleurodesis allowed. Patients who require supplemental oxygen or with oxygen saturation on room air <89% are not eligible. Pericardial effusions of any grade are not eligible.
4. Untreated documented symptomatic central nervous system (CNS) metastases.
5. Cardiac Symptoms:

   1. Uncontrolled angina, congestive heart failure(CHF)or myocardial infarction within 6 months
   2. Diagnosed congenital long QT syndrome
   3. Any h/o clinically significant ventricular arrhythmias
   4. Prolonged QT corrected (QTc) interval on pre-entry EKG (>450 msec)
   5. Uncontrolled B/P as defined as >160/90 on B/P therapy
6. Hypokalemia or hypomagnesaemia if it cannot be corrected.
7. H/o diagnosed congenital acquired bleeding disorders.
8. Ongoing or recent (≤3 months) significant (≥grade 3) GI bleeding.
9. Con Meds:

   1. Drugs having risk of causing Torsades de Pointes (must stop drug 7 days before dasatinib);
   2. Current therapeutic dose unfractionated heparin, low-molecular weight heparin, or coumadin therapy;
   3. St. John's Wort must be stopped while on dasatinib;
   4. IV bisphosphonates stopped 2 weeks pre/6 weeks post dasatinib.
10. Prisoners/subjects compulsorily detained for tx of psychiatric and/or physical illness.
11. Pregnant or breastfeeding.
12. Active or uncontrolled infection requiring IV antibiotics.
13. Impairment of GI function/disease that may alter absorption of dasatinib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
14. Received investigational drugs ≤4 weeks prior to starting study drug and/or not recovered from side effects of such therapy. Any other anti-neoplastic and/or molecular therapy must be discontinued 7 days prior to starting dasatinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kelley, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Durham VA Medical Center, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Duke Raleigh, Raleigh, North Carolina

REFERENCES:
- [Background] Downward J. Cancer biology: signatures guide drug choice. Nature. 2006 Jan 19;439(7074):274-5. doi: 10.1038/439274a. No abstract available. PMID 16421553
- See also: Clinical Trials at Duke Comprehensive Cancer Center — http://www.cancer.duke.edu/CTrials/index.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study opened to enrollment in November 2008 and closed in October 2011 due to slow accrual. Subjects were enrolled at 3 sites: Duke University Medical Center, Durham VA Medical Center, and the University of Minnesota. All subjects were enrolled in Stage 1, in which prior knowledge of each subject's tumoral Src-activity was not known.
Groups:
- Dasatinib: Dasatinib: 70 mg PO twice daily until progression.
Period: Overall Study
Arm/Group | Dasatinib
Started | 37 (Signed a consent form)
Completed | 25 (Received at least one dose of study drug)
Not Completed | 12
Not completed — Screen failure/Ineligible | 10
Not completed — No Reason Provided | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All consented subjects included in baseline analysis.
Arm/Group | Dasatinib
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: Tumor response rate was defined by RECIST criteria:
  CR (complete response) = disappearance of all target lesions taking as reference the baseline sum of the longest diameter (LD); PR (partial response) = at least a 30% decrease in the sum of the longest diameter of target lesions; PD (progressive disease) = at least a 20% increase in the sum of the longest diameter of target lesions as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; SD (stable disease) = Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as reference the smallest sum LD since the treatment started
Time Frame: 2 years
Population: Unable to determine the response for 9 subjects.
Measure: Number; unit: participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 16
participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 5
  Progression of Disease | 11

2. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is the duration from date of consent to date of death from any cause.
Time Frame: Progression and survival every 6 months
Population: All subjects who received at least one dose of dasatinib were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dasatinib
Number analyzed (Participants) | 25
months | 3.7 [2.3 to 5.9]

3. Secondary Outcome: Grade 3-5 Toxicity Associated With Dasatinib Treatment
Description: Number of subjects with Grade 3-5 toxicity as assessed using NCI CTCAE criteria with the attribution of possibly, probably, or definitely related to protocol treatment.
Time Frame: Duration of dasatinib treatment plus 30 days
Population: All subjects who received at least one dose of dasatinib were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 25
participants | 12

4. Secondary Outcome: Describe Change in Serum Levels of C-terminal Cross-linked Collagen I Between Pre-treatment and 6 Weeks After Starting Dasatinib.
Time Frame: 2 years
Population: Assays were not run because no objective tumor response was observed.
Arm/Group | Dasatinib
Number analyzed (Participants) | 0

5. Secondary Outcome: Determine Relationship Between K-ras Gene Mutation and Response to Dasatinib.
Time Frame: 2 years
Population: Assays were not run because no objective tumor response was observed.
Arm/Group | Dasatinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Evalulable Patients That Received Dasatinib: Dasatinib: 70 mg PO twice daily until progression.
Arm/Group | Evalulable Patients That Received Dasatinib
Serious Adverse Events (participants affected / at risk) | 17/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Evalulable Patients That Received Dasatinib (N=25)
anorexia (General disorders) | 1 — NCI CTCAE version 3.0
decreased hemoglobin (Blood and lymphatic system disorders) | 1 — NCI CTCAE version 3.0
decreased leukocytes (Blood and lymphatic system disorders) | 1 — NCI CTCAE version 3.0
dehydration (General disorders) | 1 — NCI CTCAE version 3.0
dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 — NCI CTCAE version 3.0
fatigue (General disorders) | 5 — NCI CTCAE version 3.0
hyponatremia - metabolic/lab (General disorders) | 1 — NCI CTCAE version 3.0
muscle weakness (generalized) (General disorders) | 1 — NCI CTCAE version 3.0
nausea (Gastrointestinal disorders) | 2 — NCI CTCAE version 3.0
neuro-motor (generalized weakness) (General disorders) | 1 — NCI CTCAE version 3.0
pericardial effusion (General disorders) | 1 — NCI CTCAE version 3.0
vomiting (Gastrointestinal disorders) | 1 — NCI CTCAE version 3.0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Evalulable Patients That Received Dasatinib (N=25)
anorexia (General disorders) | 6 — NCI CTCAE version 3.0
bronchospasm (wheezing) (Respiratory, thoracic and mediastinal disorders) | 2 — NCI CTCAE version 3.0
decreased hemoglobin (Blood and lymphatic system disorders) | 8 — NCI CTCAE version 3.0
decreased neutrophils (Blood and lymphatic system disorders) | 1 — NCI CTCAE version 3.0
diarrhea (Gastrointestinal disorders) | 3 — NCI CTCAE version 3.0
dizziness (lightheadedness) (General disorders) | 1 — NCI CTCAE version 3.0
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 — NCI CTCAE version 3.0
edema (periorbital/face) (General disorders) | 1 — NCI CTCAE version 3.0
elevated AST (Blood and lymphatic system disorders) | 2 — NCI CTCAE version 3.0
elevated creatinine (Renal and urinary disorders) | 1 — NCI CTCAE version 3.0
elevated LDH (General disorders) | 1 — NCI CTCAE version 3.0
fatigue (General disorders) | 8 — NCI CTCAE version 3.0
flatulence (Gastrointestinal disorders) | 1 — NCI CTCAE version 3.0
hair loss (alopecia) (Skin and subcutaneous tissue disorders) | 1 — NCI CTCAE version 3.0
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 — NCI CTCAE version 3.0
insomnia (General disorders) | 1 — NCI CTCAE version 3.0
leukocytosis (General disorders) | 1 — NCI CTCAE version 3.0
muscle weakness - lower extremity (leg weakness) (General disorders) | 1 — NCI CTCAE version 3.0
muscle weakness (generalized) (General disorders) | 1 — NCI CTCAE version 3.0
myalgias (generalized) (Musculoskeletal and connective tissue disorders) | 1 — NCI CTCAE version 3.0
nausea (Gastrointestinal disorders) | 6 — NCI CTCAE version 3.0
neutrophils (neutropenia) (Blood and lymphatic system disorders) | 1 — NCI CTCAE version 3.0
pain extremity (legs) (General disorders) | 1 — NCI CTCAE version 3.0
pain-joint (Musculoskeletal and connective tissue disorders) | 1 — NCI CTCAE version 3.0
pedal edema (General disorders) | 1 — NCI CTCAE version 3.0
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 — NCI CTCAE version 3.0
pleural effusion, bilateral (Respiratory, thoracic and mediastinal disorders) | 1 — NCI CTCAE version 3.0
pulmonary edema (Cardiac disorders) | 1 — NCI CTCAE version 3.0
rash (Skin and subcutaneous tissue disorders) | 6 — NCI CTCAE version 3.0
renal/genitourinary other (slow starting urinary stream) (Renal and urinary disorders) | 1 — NCI CTCAE version 3.0
taste alteration (Gastrointestinal disorders) | 3 — NCI CTCAE version 3.0
ulcers (scrotal) (Skin and subcutaneous tissue disorders) | 1 — NCI CTCAE version 3.0
vomiting (Gastrointestinal disorders) | 2 — NCI CTCAE version 3.0
weight loss (General disorders) | 2 — NCI CTCAE version 3.0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes